CLINICAL TRIAL: NCT01727895
Title: Effects of Orally Administered Beta-glucan on Leukocyte Function in Humans, a Pilot Study
Brief Title: Effects of Orally Administered Beta-glucan on Leukocyte Function in Humans
Acronym: BG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Betaglucan_immunity
Record Dates: First submitted 2012-11-12; First posted 2012-11-16 (Estimated); Results first posted 2014-07-31 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Immunologic Deficiency Syndromes
Keywords: Betaglucan, immune modulation, immunoparalysis, immune suppression
MeSH Terms: conditions — Immunologic Deficiency Syndromes | interventions — beta-Glucans

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Beta-glucan (Experimental): Commercial available Beta-glucan derived from bakers yeast (S. Cerevisiae): Glucan #300® produced by Transferpoint, Columbia, United States. 2 capsules of 500mg Glucan #300®, daily, for seven days.
  Interventions: Dietary Supplement: Beta-glucan (Glucan #300®)
- Control group (No Intervention)

INTERVENTIONS:
Dietary Supplement: Beta-glucan (Glucan #300®)
  Arms: Beta-glucan

SUMMARY:
The purpose of this study is to test wether orally administered Beta-glucan has systemic effects in humans.

DETAILED DESCRIPTION:
The immunostimulatory properties of mushrooms have been recognized for centuries, and "medicinal" mushrooms are still widely used in alternative medicine all over the world. Although a number of fungal components have been implicated in these properties, Beta-glucans have attracted the most attention. However, although Beta-glucans are widely used as a health food supplement, their immunomodulatory effects after administration in humans have not yet been determined.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥18
* Healthy males

Exclusion Criteria:

* Subjects with a history of allergy or intolerance to Beta-glucan
* Use of any medication
* Participation in a drug trial or donation of blood 3 months prior to Beta-glucan administration
* Use of antibiotics, norit, laxatives (up till 6 months prior to inclusion), cholestyramine, acid burn inhibitors or immune suppressive agents (up till 3 months prior to inclusion), and pre- and probiotics (up till 1 month prior to inclusion).

Ages: 18 Years to 36 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Netea, MD, PhD, Principal Investigator — Radboud University Nijmegen Medical Centre, The Netherlands
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] Leentjens J, Quintin J, Gerretsen J, Kox M, Pickkers P, Netea MG. The effects of orally administered Beta-glucan on innate immune responses in humans, a randomized open-label intervention pilot-study. PLoS One. 2014 Sep 30;9(9):e108794. doi: 10.1371/journal.pone.0108794. eCollection 2014. PMID 25268806

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from April until May 2013 in the Radboud University Medical Centre Nijmegen.
Pre-assignment Details: Exclusion of subjects was based on pre-defined exclusion criteria or the unability of subjects to comply with the study time schedule.
Groups:
- Beta-glucan: Commercial available Beta-glucan derived from bakers yeast (S. Cerevisiae): Glucan #300® produced by Transferpoint, Columbia, United States. 2 capsules of 500mg Glucan #300®, daily, for seven days.
  Beta-glucan (Glucan #300®)
- Control Group: No intervention
Period: Overall Study
Arm/Group | Beta-glucan | Control Group
Started | 10 | 5
Completed | 10 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Beta-glucan | Control Group | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 20 [19 to 22] | 20 [19 to 24] | 20 [19 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 5 | 15
TNF-α Secretion by ex Vivo LPS-Stimulated Peripheral Blood mononuclear cells [Median (Inter-Quartile Range); unit: pg/ml] | 691 [276 to 2649] | 749 [287 to 1160] | 720 [282 to 1905]

OUTCOME MEASURES:

1. Primary Outcome: Tumor Necrosis Factor (TNF)-α Secretion by ex Vivo Lipopolysaccharide (LPS)-Stimulated Peripheral Blood Mononuclear Cells (PBMCs)
Description: The primary objective of the study is to evaluate the systemic effects of orally administered Beta-glucan on innate immune responses of leukocytes. The effects of Beta-glucan will be determined by measuring the ex vivo responsiveness of leukocytes to various inflammatory stimuli as a surrogate marker of the antimicrobial response
Time Frame: up to 21 days
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Beta-glucan | Control Group
Number analyzed (Participants) | 10 | 5
pg/ml | 691 [276 to 2649] | 749 [287 to 1160]

2. Secondary Outcome: • Production of Other Cytokines (TNF-α, Interleukin (IL)-6, IL-10, IL-1β, IL-17, IL-22, Interferon (IFN)-γ) by Leukocytes ex Vivo Stimulated With Various Stimuli (Including LPS, Pam3Cys, Mycobacterium Tuberculosis, Poly(I:C), Candida, Staph Aureus)
Time Frame: days 0, 6, 21
Reporting Status: Not Posted

3. Secondary Outcome: • the Absorbance of Orally Administered Beta-glucan Into the Blood Compartment, Measured by ELISA
Time Frame: Days 0, 6, 21
Reporting Status: Not Posted

4. Secondary Outcome: • Transcriptional Pathways (by Use of Microarrays) With Focus on Inflammatory Pathways.
Time Frame: Days 0, 6, 21
Reporting Status: Not Posted

5. Secondary Outcome: • Changes in Phenotype and Gene Expression Caused by Mechanisms Other Than Changes in the Underlying DNA Sequence (Epigenetic Modifications)
Time Frame: Days 0, 6, 21
Reporting Status: Not Posted

6. Secondary Outcome: • the Leukocyte Capacity to Phagocytose and Kill the Fungal Pathogen Candida Albicans (Antifungal Activity).
Time Frame: Days 0, 6, 21
Reporting Status: Not Posted

7. Secondary Outcome: the Composition of Faecal Microbiota
Time Frame: Days 0, 6, 21
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Beta-glucan | Control Group
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 1/10 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Beta-glucan (N=10) | Control Group (N=5)
Flare of acne, one week after discontinuation of Beta-glucan intake (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes